CLINICAL TRIAL: NCT03230058
Title: Combination Treatment of 5% Natamycin and 1% Voriconazole in Fungal Keratitis: a Prospective Randomized Double Masked Clinical Trial
Brief Title: Combination Treatment of 5% Natamycin and 1% Voriconazole in Fungal Keratitis
Acronym: NATA_VORI
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: L.V. Prasad Eye Institute (Other)
Responsible Party: Principal Investigator, Charitha, MS, L.V. Prasad Eye Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GMRV_NATA01
Record Dates: First submitted 2017-07-23; First posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Infection, Fungal
MeSH Terms: conditions — Mycoses | interventions — Suspensions; Voriconazole; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 (Experimental): Once the patient is randomized to either of the 2 groups using computer-generated randomization blocks, the hospital pharmacist would provide the appropriate medications. The treating ophthalmologist, microbiologist and patients will be masked to the drug by using similar vials. The experimental group (Group 1) will receive 1% voriconazole eye drop (Aurolab, Madurai, India) + 5% Natamycin ophthalmic suspension eye drop hourly (USP 5% Natamet, M.J. Pharmaceuticals, Mumbai, India).
  The subjects will be hospitalized for at least 4 days with medications given by the ward nurse.
  Patients will be followed up every week after being discharged until complete resolution is noted.
  Interventions: Drug: Group 1 Natamycin 5% Suspension + voriconazole 1% eye drops; Group 2 Natamycin 5% Suspension + Vehicle eye drops
- group 2 (Placebo Comparator): Once the patient is randomized to either of the 2 groups using computer-generated randomization blocks, the hospital pharmacist would provide the appropriate medications. The treating ophthalmologist, microbiologist and patients will be masked to the drug by using similar vials. The placebo group (Group 2) will receive Vehicle eye drops + 5% Natamycin ophthalmic suspension every hour (USP 5% Natamet, M.J. Pharmaceuticals, Mumbai, India).
  The subjects will be hospitalized for at least 4 days with medications given by the ward nurse.
  Patients will be followed up every week after being discharged until complete resolution is noted.
  Interventions: Drug: Group 1 Natamycin 5% Suspension + voriconazole 1% eye drops; Group 2 Natamycin 5% Suspension + Vehicle eye drops

INTERVENTIONS:
Drug: Group 1 Natamycin 5% Suspension + voriconazole 1% eye drops; Group 2 Natamycin 5% Suspension + Vehicle eye drops — instillation of drops

SUMMARY:
OBJECTIVE To evaluate the efficacy and safety of the concurrent treatment of 5% Natamycin and 1% Voriconazole in patients affected by fungal keratitis METHODS AND MATERIALS STUDY POPULATION Patients with smear and or culture proven fungal keratitis presenting to our Instituts, were eligible for enrollment.

STUDY DESIGN Prospective double masked randomized clinical trial.

DETAILED DESCRIPTION:
PROTOCOL FOR SUBMISSION AND APPROVAL OF RESEARCH PROJECT

TITLE:

Combination treatment of 5% Natamycin and 1% Voriconazole in fungal keratitis: a Prospective Randomized double masked clinical trial STUDY LOCATION LV Prasad Eye Institute, GMR Varalakshmi Campus, Visakhapatnam, Andhra Pradesh, India INVESTIGATORS Dr Merle Fernandes Consultant, Cornea and Anterior Segment Service LV Prasad Eye Institute, GMR Varalakshmi Campus Visakhapatnam, Andhra Pradesh, India Dr Antonio Di Zazzo Fellow, Cornea and Anterior Segment Service LV Prasad Eye Institute, GMR Varalakshmi Campus Visakhapatnam, Andhra Pradesh, India

Dr J V Raghava Consultant, Cornea and Anterior Segment Service LV Prasad Eye Institute, GMR Varalakshmi Campus Visakhapatnam, Andhra Pradesh, India

Dr Sayali Sane Fellow, Cornea and Anterior Segment Service LV Prasad Eye Institute, GMR Varalakshmi Campus Visakhapatnam, Andhra Pradesh, India

Dr Siddarth Yadav Fellow, Cornea and Anterior Segment Service LV Prasad Eye Institute, GMR Varalakshmi Campus Visakhapatnam, Andhra Pradesh, India

INTRODUCTION Fungal Keratitis Microbial keratitis is a leading cause of monocular blindness worldwide, being second only to cataract as per WHO bulletin.[1]Fungal keratitis represents almost half of all cases of suppurative keratitis in some parts of the developing world[2] and comprises 30-40% of all cases of culture-positive infectious keratitis particularly in South India[3, 4]. Filamentous fungi have been reported as causative agents in large proportions of mycotic corneal ulcers in tropical climates as compared to temperate climates[1].

Despite high prevalence of fungal keratitis, the treatment of fungal keratitis is more challenging than bacterial keratitis for several reasons including but not limited to the following: few commercially available topical anti-fungal agents, fungistatic drugs, limited ocular penetration, insubstantial research and development into newer agents. , Studies of longer duration elucidate that monocular vision loss from fungal corneal ulcers had an impact on psychosocial functioning apart from its effect on mobility and activity limitation, especially among those with severe vision loss in the involved eye.[5, 6] In addition it has been well established that poor vision is associated with depression. [7] Current treatment for fungal keratitis Few published randomized controlled trial compare alternative antifungal therapy for mycotic keratitis[8, 9], and no new ocular antifungal medications have been approved by the Food and Drug Administration since amphotericin B and natamycin were approved in the 1960s [10].

Currently, fungal infections of the cornea are difficult to eradicate as fungi often resist treatment. Management of fungal keratitis requires timely diagnosis of the infection and administration of appropriate antifungal therapy. Antifungal agents are still the major therapeutic options in fungal keratitis, whereby success depends on the agent's ability to penetrate into the aqueous and achieve therapeutic levels [11].

Natamycin Natamycin, the only FDA-approved agent for the treatment of fungal keratitis, is a fungicidal tetraene polyene antibiotic, derived from Streptomyces natalensis that possesses in vitro activity against a variety of yeast and filamentous fungi, including Candida, Aspergillus, Cephalosporium, Fusarium and Penicillium species[12]. Therefore Natamycin is the preferred drug of choice for filamentous fungal keratitis. Topical Natamycin poorly penetrates an intact epithelium and often requires manual debridement of the corneal epithelium for greater efficacy. It has a antimicrobial power as effective as Econazole[8], more effective than Itraconazole[13], and more rapidly acting than Terbinafine[14],. Topical Natamycin has been superior to topical Voriconazole for the treatment of filamentous fungal corneal ulcers, and in particular those culture-positive for Fusarium species [15, 16].

Voriconazole Newer triazoles (Voriconazole, Posaconazole and Ravuconazole) have been suggested as better alternatives in the treatment of fungal keratitis not responding to conventional antifungals. They are fungistatic and act by inhibiting biosynthesis of ergosterol, an essential component in fungal cell wall[17]. Voriconazole is active against both filamentous fungi and Candida species and has recently become the treatment of choice for systemic diseases such as pulmonary aspergillosis[18]. Numerous case reports in the ophthalmic literature have described the use of Voriconazole in fungal keratitis [17, 19-24]. The superiority of these agents compared with natamycin has not been established Topical voriconazole has good penetration into the eye (0.61-3.30 mg/L in the aqueous humor after 1 h of topical administration)[25]. Recent randomized controls have not reported greater efficacy of 1% voriconazole, (reconstituted from injection vial) compared to 5% natamycin eye drops (imported from USA) in fungal keratitis[16, 26].

While Natamycin is a good drug to treat fungal keratitis, but treatment failures have been reported by several authors[27]. Natamycin has been reported as the most effective medication against filamentous fungi, but large ulcer size, hypopyon and Aspergillus as causative organism have been reported as predictors of poor outcome with topical 5% natamycin monotherapy [28]. The search for a better broad spectrum antifungal drug to treat fungal keratitis continues. There have been studies using a combination of antifungal agents, in order to develop a multidrug therapy[ 29, 30]. Amphoptericin B and Flucytosine have been described to have synergistic effects.15 while Natamycin and Etoconazole have also been used effectively in an animal model of Aspergillus keratitis[18]. A randomized clinical trial testing efficacy of 2% Econazole as a topical preparation added to 5% Natamycin for the treatment of fungal keratitis in south India[2, 8]did not show any advantage compared to monotherapy with Natamycin [2] .A combination of a Polyene (Amphotericin B) and a triazole (Voriconazole) is synergistic at low median concentrations when tested against Aspergillus species in vitro, suggesting a concentration dependent interaction between the 2 drug.[31].

The efficacy of a concurrent therapy with Natamycin and Voriconazole has been not been systematically studied, as well as the potential synergistic effect this combination could have on the management of fungal corneal infection.

OBJECTIVE To evaluate the efficacy and safety of the concurrent treatment of 5% Natamycin and 1% Voriconazole in patients affected by fungal keratitis METHODS AND MATERIALS STUDY POPULATION Patients with smear and or culture proven fungal keratitis presenting to our Instituts, were eligible for enrollment.

STUDY DESIGN Prospective double masked randomized clinical trial. The subject will be enrolled in 2 groups of 20 subjects each. The first group will start on concurrent topical treatment of 5% Natamycin and 1% Voriconazole hourly, the second group will start on concurrent topical treatment of 5% Natamycin and placebo (Voriconazole vehicle) one hourly. All patients will also be started on topical cycloplegics, oral Ketoconazole and oral non steroidal anti inflammatory agents and anti glaucoma medications when necessary.

Inclusion Criteria Subjects > 18 yrs of age Willing to give appropriate informed consent Presence of corneal ulcer measuring > 2mm in vertical and horizontal dimensions at presentation (epithelial defect and signs of stromal inflammation) Microbiologic evidence of fungus on smear and or culture media Willing to return for all the follow up visits Exclusion Criteria Patients not willing to give consent Patients unable to cooperate for the procedure Patient with impending, or actual perforation or bilateral corneal ulcer or scleral involvement History of previous ocular surgery Evidence of bacterial, parasitic or viral infection or co-infection Previous corneal scar Known allergy to the study medication (drug or preservative) Pregnant or nursing females Immunocompromised patients

END POINTS

Definitions

Ulcer Healing, resolving keratitis or worsening keratitis:

An ulcer will be defined healed if the ulcer heals with formation of a corneal scar Lesion will be classified as resolving keratitis if the corneal infiltrate reduces in size by at least 1 mm and or decrease in endothelial plaque or satellite lesions, appearance of scarring, accompanied by reduction in symptoms An ulcer will be deemed to demonstrate no response or worsening when it will show a lack of improvement or worsening in inflammatory sign scores or stromal infiltrate dimensions or corneal melt and deterioration in any clinical examination factor.

Primary End point:

Complete success: Complete resolution of the infiltrate with formation of a scar on medical treatment alone Partial success: Complete resolution of the infiltrate on medical treatment and use of cyanoacrylate glue and bandage contact lens Failure: Worsening of the ulcer necessitating therapeutic penetrating keratoplasty of evisceration

Secondary Endpoint:

Best-corrected visual acuity (logarithm of the minimum angle of resolution (logMAR)).

Evidence of ocular surface toxic reaction assessed by follicular reaction in the lower forniceal conjunctiva, superficial punctate keratopathy, congestion in the lower bulbar conjunctiva

CONSENT All subjects will give informed consent before participating. The research protocol will adhere to the tenets of the Declaration of Helsinki.

PROCEDURE Patients will be selected from the out-patient department and screened for entry into the study. 20 Subjects will be randomized to Natamycin+Voriconazole and 20 to Natamycin +Vehicle using a computer assisted random number generato (Appendix 1).

All subjects will undergo a detailed history, refraction, unaided and best corrected LogMAR visual acuity recording, applanation tonometry in the unaffected eye, slit lamp biomicroscopic evaluation and measurement of the epithelial defect and ulcer along maximum length and perpendicular to this along the maximum width, percentage of thinning, depth of the infiltrate, presence of satellite lesions, endothelial exudates, height of hypopyon and indirect ophthalmoscopy or ultrasound biomicroscopy for fundus evaluation, wherever needed.

The details regarding the symptoms associated with the corneal ulcer, its onset, duration and progression, and history of predisposing factors such as trauma, steroid use, use of bandage contact lens, pre-existing ocular surface disorder and diabetes will be also elicited.

All patients microbial keratitis will undergo a detailed microbiological evaluation with a corneal scraping using a #15 blade for Gram stain and 10% potassium hydroxide -calcofluor white wet mount and subsequently plated for cultures (blood agar, chocolate agar, Saboraud's dextrose agar, potato dextrose agar. non-nutrient agar, thioglycollate broth, brain heart infusion broth.

RANDOMIZATION, ALLOCATION CONCEALMENT AND ADMINISTRATION OF MEDICATION Once the patient is randomized to either of the 2 groups using computer-generated randomization blocks, the hospital pharmacist would provide the appropriate medications. The treating ophthalmologist, microbiologist and patients will be masked to the drug by using similar vials. One group will receive 1% voriconazole eye drop (Aurolab, Madurai, India) + 5% Natamycin ophthalmic suspension eye drop hourly and the other group receiving Vehicle eye drops+ 5% Natamycin ophthalmic suspension every hour (USP 5% Natamet, M.J. Pharmaceuticals, Mumbai, India).

The subjects will be hospitalized for at least 2 weeks with medications given by the ward nurse.

Patients will be followed up every week after being discharged until complete resolution is noted.

SLIT LAMP PHOTOGRAPHY Slit lamp photographs will be taken at presentation and weekly intervals until complete resolution.

MICROBIOLOGICAL EXAMINATION Corneal scrapings will be collected using blade no.15, under topical anaesthesia at the slit lamp as per our Institute protocol described earlier. (Ref). The slides will be stained with Gram stain and 10% potassium hydroxide with 0.1% calcofluor white wet mount for direct microscopy. Corneal scrapings will be inoculated in the following culture media : BA, CA, PDA, SDA, BHI, thioglyocollate, NNA. All media will be held for 2 weeks in case of no growth before declaring the sample as sterile.

How often and how they will be selected?

Patients will be selected from the out-patient department and screened for entry into the study. Sample size of 40 subjects will be selected with 20 subjects in each age group

How often and how many will be studied? Sample size of 40 subjects will be selected with 20 subjects in each age group, until complete resolution of the infiltrate. The follow up visits will be based on clinical condition.

Which consultant(s) will be responsible for the patients? All cornea consultants of LVPEI GMR Varalakshmi campus will be responsible for the subjects.

Normal volunteers - From where will they be recruited? How many? Not applicable

At the time of their participation in the study, will the subjects be involved in any other experimental work? Please give details.

NO

List the exact procedures and how often the subjects will be submitted to such procedures, i.e collection of urine and faeces, vene-puncture, intubation, special diet, drugs administered with dose excluding radio-isotopes or irradiation.

Complete eye examination Microbiological assessment(as needed, at screening visit) Slit lamp Photography Drug administration (5% Natamycin ophthalmic suspension eye drops, 1% Voriconazole eye drops, every hour, daily) State any potential or known hazards of the procedures listed above. How does the investigator intend to overcome these? N/A

Give any details of any procedures involving radio-isotopes or irradiation. N/A

What is the investigator's personal experience with the proposed technique? Good N/A How will the informed consent be taken and by whom? The consent will be taken by the participating investigators and their counselors.

Please details whether the subjects are to be reimbursed expensed incurred during participation in the study and also whether or not it is contemplated giving them a gift or token of any sort. If so, please state the exact amount.

NA

Is the protocol, copy of the patient's information and consent form appended with the application.

Yes

Action plan for reporting adverse reaction to Ethics Committee and other participants of the study.

Ethics committee meetings are held every month. Adverse events will be recorded in the Incident report form and also in the CRF (clinical research file). The information will be presented to the faculty member who is part of the EC and will be presented to the EC at the next meeting.

Outcome measures: Complete resolution of infiltrate resulting in scar formation

Any other information that you would like to provide to the Ethics Committee. No

Signatures of the Investigators and Co-investigators.

REFERENCES

1. Srinivasan, M., Fungal keratitis. Curr Opin Ophthalmol, 2004. 15(4): p. 321-7.
2. Prajna, N.V., et al., Concurrent use of 5% natamycin and 2% econazole for the management of fungal keratitis. Cornea, 2004. 23(8): p. 793-6.
3. Bharathi, M.J., et al., Epidemiological characteristics and laboratory diagnosis of fungal keratitis. A three-year study. Indian J Ophthalmol, 2003. 51(4): p. 315-21.
4. Chowdhary, A. and K. Singh, Spectrum of fungal keratitis in North India. Cornea, 2005. 24(1): p. 8-15.
5. Mathews, P.M., et al., Severity of vision loss interacts with word-specific features to impact out-loud reading in glaucoma. Invest Ophthalmol Vis Sci, 2015. 56(3): p. 1537-45.
6. Finger, R.P., et al., The impact of the severity of vision loss on vision-specific functioning in a German outpatient population - an observational study. Graefes Arch Clin Exp Ophthalmol, 2011. 249(8): p. 1245-53.
7. Qian, Y., et al., Depression and visual functioning in patients with ocular inflammatory disease. Am J Ophthalmol, 2012. 153(2): p. 370-378 e2.
8. Prajna, N.V., et al., A randomised clinical trial comparing 2% econazole and 5% natamycin for the treatment of fungal keratitis. Br J Ophthalmol, 2003. 87(10): p. 1235-7.
9. Sharma, S., et al., Re-appraisal of topical 1% voriconazole and 5% natamycin in the treatment of fungal keratitis in a randomised trial. Br J Ophthalmol, 2015. 99(9): p. 1190-5.
10. Whitcher, J.P., M. Srinivasan, and M.P. Upadhyay, Corneal blindness: a global perspective. Bull World Health Organ, 2001. 79(3): p. 214-21.
11. Manzouri, B., G.C. Vafidis, and R.K. Wyse, Pharmacotherapy of fungal eye infections. Expert Opin Pharmacother, 2001. 2(11): p. 1849-57.
12. O'Day, D.M., Selection of appropriate antifungal therapy. Cornea, 1987. 6(4): p. 238-45.
13. Kalavathy, C.M., et al., Comparison of topical itraconazole 1% with topical natamycin 5% for the treatment of filamentous fungal keratitis. Cornea, 2005. 24(4): p. 449-52.
14. Liang, Q.F., et al., Effect of topical application of terbinafine on fungal keratitis. Chin Med J (Engl), 2009. 122(16): p. 1884-8.
15. Rose-Nussbaumer, J., et al., Risk factors for low vision related functioning in the Mycotic Ulcer Treatment Trial: a randomised trial comparing natamycin with voriconazole. Br J Ophthalmol, 2015.
16. Prajna, N.V., et al., The mycotic ulcer treatment trial: a randomized trial comparing natamycin vs voriconazole. JAMA Ophthalmol, 2013. 131(4): p. 422-9.
17. Kofla, G. and M. Ruhnke, Voriconazole: review of a broad spectrum triazole antifungal agent. Expert Opin Pharmacother, 2005. 6(7): p. 1215-29.
18. Komadina, T.G., et al., Treatment of Aspergillus fumigatus keratitis in rabbits with oral and topical ketoconazole. Am J Ophthalmol, 1985. 99(4): p. 476-9.
19. Creti, A., et al., Voriconazole curative treatment for Acremonium species keratitis developed in a patient with concomitant Staphylococcus aureus corneal infection: a case report. In Vivo, 2006. 20(1): p. 169-71.
20. Ozbek, Z., et al., Voriconazole in the management of Alternaria keratitis. Cornea, 2006. 25(2): p. 242-4.
21. Bernal, M.D., et al., Outbreak of Fusarium keratitis in soft contact lens wearers in San Francisco. Arch Ophthalmol, 2006. 124(7): p. 1051-3.
22. Klont, R.R., et al., Successful treatment of Fusarium keratitis with cornea transplantation and topical and systemic voriconazole. Clin Infect Dis, 2005. 40(12): p. e110-2.
23. Dupuis, A., et al., Preparation and stability of voriconazole eye drop solution. Antimicrob Agents Chemother, 2009. 53(2): p. 798-9.
24. Hariprasad, S.M., et al., Voriconazole in the treatment of fungal eye infections: a review of current literature. Br J Ophthalmol, 2008. 92(7): p. 871-8.
25. Thiel, M.A., et al., Voriconazole concentration in human aqueous humor and plasma during topical or combined topical and systemic administration for fungal keratitis. Antimicrob Agents Chemother, 2007. 51(1): p. 239-44.
26. Prajna, N.V., et al., Comparison of natamycin and voriconazole for the treatment of fungal keratitis. Arch Ophthalmol, 2010. 128(6): p. 672-8.
27. FlorCruz, N.V. and J.R. Evans, Medical interventions for fungal keratitis. Cochrane Database Syst Rev, 2015. 4: p. CD004241.
28. Lalitha, P., et al., Risk factors for treatment outcome in fungal keratitis. Ophthalmology, 2006. 113(4): p. 526-30.
29. Lee, S.J., J.J. Lee, and S.D. Kim, Topical and oral voriconazole in the treatment of fungal keratitis. Korean J Ophthalmol, 2009. 23(1): p. 46-8.
30. Bunya, V.Y., et al., Topical and oral voriconazole in the treatment of fungal keratitis. Am J Ophthalmol, 2007. 143(1): p. 151-3.
31. O'Shaughnessy, E.M., et al., Antifungal interactions within the triple combination of amphotericin B, caspofungin and voriconazole against Aspergillus species. J Antimicrob Chemother, 2006. 58(6): p. 1168-76.

POWER CALCULATION:

α = level of significance(0.05)

1-β = power of the test(80%) σ = standard deviation (9%, assumed) ε= clinically meaningful difference (5%, assumed) Total Sample size 50 + 10% lost to follow(5)=55 The required sample size to achieve an 80% power at 5% level of significance for detecting clinically meaningful difference (suppose a difference of 5% in healing is considered of clinically meaningful difference) with assuming that the standard deviation is 9%,is 55 for each group(Gr1 Nata + placebo=55, Gr2 Nata + Vori =55).

Statistical Test to be used for analyzing the results: Exploratory data analysis (EDA), ANOVA, T-test, linear Mixed effect models.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 18 yrs of age Willing to give appropriate informed consent Presence of corneal ulcer measuring > 2mm in vertical and horizontal dimensions at presentation (epithelial defect and signs of stromal inflammation) Microbiologic evidence of fungus on smear and or culture media Willing to return for all the follow up visits

Exclusion Criteria:

* Patients not willing to give consent Patients unable to cooperate for the procedure Patient with impending, or actual perforation or bilateral corneal ulcer or scleral involvement History of previous ocular surgery Evidence of bacterial, parasitic or viral infection or co-infection Previous corneal scar Known allergy to the study medication (drug or preservative) Pregnant or nursing females Immunocompromised patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Success or failure | 8 weeks
  Primary End point:
  Complete success: Complete resolution of the infiltrate with formation of a scar on medical treatment alone Partial success: Complete resolution of the infiltrate on medical treatment and use of cyanoacrylate glue and bandage contact lens Failure: Worsening of the ulcer necessitating therapeutic penetrating keratoplasty or evisceration

SECONDARY OUTCOMES:
Best-corrected visual acuity | 8 weeks
  improvement in best corrected visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: merle fernandes, MS, Principal Investigator — LVPEI
Locations (1):
- GMRV Campus LV Prasad Eye Insitute, Visakhapatnam, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sharma S, Das S, Virdi A, Fernandes M, Sahu SK, Kumar Koday N, Ali MH, Garg P, Motukupally SR. Re-appraisal of topical 1% voriconazole and 5% natamycin in the treatment of fungal keratitis in a randomised trial. Br J Ophthalmol. 2015 Sep;99(9):1190-5. doi: 10.1136/bjophthalmol-2014-306485. Epub 2015 Mar 4. PMID 25740805
- [Result] Srinivasan M. Fungal keratitis. Curr Opin Ophthalmol. 2004 Aug;15(4):321-7. doi: 10.1097/00055735-200408000-00008. PMID 15232472
- [Derived] Di Zazzo A, Surico PL, Parmar UPS, Tarini S, De Luca A, Madduri B, Mohan N, Fernandes M. Efficacy of natamycin monotherapy versus combination therapy with voriconazole for fungal keratitis: a randomised clinical trial. Br J Ophthalmol. 2025 Dec 9:bjo-2025-328695. doi: 10.1136/bjo-2025-328695. Online ahead of print. PMID 41365527